MEDICAL RECORD

## CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

• Adult Patient or

• Parent, for Minor Patient

INSTITUTE: National Cancer Institute

STUDY NUMBER: 13-C-0016 PRINCIPAL INVESTIGATOR: Hoyoung Maeng, M.D.

STUDY TITLE: A Phase I Study of an Adenoviral Transduced Autologous Dendritic Cell Vaccine

Expressing Human HER2/neu ECTM in Adults with Tumors with 1-3+ HER2/neu

Expression

Continuing Review Approved by the IRB on 11/05/18

Amendment Approved by the IRB on 08/19/19 (O)

Date posted to web: 08/24/19

Addendum to 13-C-0016

This addendum provides new information about the study "A Phase I Study of an Adenoviral Transduced Autologous Dendritic Cell Vaccine Expressing Human HER2/neu ECTM in Adults with Tumors with 1-3+ HER2/neu Expression" on which you are enrolled. The information in the consent you signed previously is unchanged.

The NIH Clinical Center Pharmaceutical Development Service (PDS) helps to make the AdHER2 DC vaccine used in this study. The PDS was recently closed down by NIH leadership after a vial of contaminated material was discovered on another study just before it was supposed to be given to a research participant. The PDS is undergoing a full review and changes are being made to make sure that processes are in place to prevent anything like this from happening again. The FDA and NIH decided that it might be better and safer to make an exception to the PDS shutdown for some research studies as long as those decisions are made on a case by case or protocol by protocol basis. The AdHER2 DC vaccine received one of those exceptions because the parts of the vaccine made by the PDS are just used in the preparation of the vaccine and are never actually given to you, the research participant. Additionally, all of the materials used in making the AdHER2 DC vaccine have to pass many tests or they can't be used. Before giving the exception, the FDA and NIH determined that the risk to you from receiving a vaccine that includes the portions made by the PDS, before all of the reviews and changes to the PDS are finished, is extremely low.

PATIENT IDENTIFICATION

## CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

• Parent, for Minor Patient

• Adult Patient or NIH-2514-1 (07-09) P.A.: 09-25-0099

File in Section 4: Protocol Consent (2)

MEDICAL RECORD

## CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

• Adult Patient or

• Parent, for Minor Patient

STUDY NUMBER: 13-C-0016 CONTINUATION: page 2 of 2 pages

| COMPLETE APPROPRIATE ITEM(S) BELOW: | | | |
|---|---|---|---|
| A. Adult Patient's Consent | | B. Parent's Permission for Minor Patient. | |
| I have read the explanation about this study | | I have read the explanation about this study | |
| and have been given the opportunity to discuss | | and have been given the opportunity to discuss | |
| it and to ask questions. I hereby consent to | | it and to ask questions. I hereby give | |
| take part in this study. | | permission for my child to take part in this | |
| | | study. | |
| | | (Attach NIH 2514-2, Minor's Ass | ent, if |
| | | applicable.) | |
| Signature of Adult Patient/ | Date | Signature of Parent(s)/ Guardian | Date |
| Legal Representative | | | |
| Print Name | | Print Name | |
| C. Child's Verbal Assent (If Ap | plicable) | | |
| , - | • / | escribed to my child and my ch | ild agrees to |
| participate in the study. | | | _ |
| Signature of Parent(s)/Guardian Date | | Print Name | |
| . , | | | |
| | | IAS BEEN APPROVED FOR US | |
| FROM NOVEMBER | X 05, 2018 11 | HROUGH NOVEMBER 12, 2019 | • |
| Signature of Investigator | Date | Signature of Witness | Date |
| Print Name | | Print Name | |
| ·-=== - | | | |

PATIENT IDENTIFICATION

## CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY (Continuation Sheet)

• Adult Patient or

• Parent, for Minor Patient

NIH-2514-1 (07-09) P.A.: 09-25-0099

File in Section 4: Protocol Consent